CLINICAL TRIAL: NCT05899985
Title: Magnetic Sentinel Lymph Node Mapping in Upper Gastro-Intestinal Cancer: A Feasibility Clinical Investigation
Acronym: MAGMAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ferronova Pty Ltd (Industry)
Collaborators: Royal Adelaide Hospital (Other); Austin Health (Other Government); Flinders Medical Centre (Other Government); Peter MacCallum Cancer Centre, Australia (Other); South Australian Health and Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMF-3
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Gastric Cancer; Esophageal Cancer
Keywords: Sentinel lymph node
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Multi-centre, partially blinded, side-by-side comparator study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): Eligible subjects will undergo their normal standard of care treatment pathway with the added interventions described below.
  Interventions: Combination Product: FerroTrace® and FerroMag Sentinel Lymph Node Mapping (SLNM) System

INTERVENTIONS:
Combination Product: FerroTrace® and FerroMag Sentinel Lymph Node Mapping (SLNM) System — FerroTrace will be injected peri-tumorally during the surgeons staging endoscopy, with an MRI conducted 12h to 28 days after injection. The MRI will be blinded to the clinical team and will assess the location of the primary draining lymph nodes (sentinel lymph nodes or SLNs).
  Patients will proceed to standard of care neoadjuvant therapy and/or surgery. During surgery, indocyanine green (ICG) will be used to identify draining lymph nodes. Following surgery, pathologists will use FerroMag to identify SLNs which will undergo standard H&E assessment, and if negative ultras-staging (fine serial slice and immunochemistry).

SUMMARY:
This is a multi-centre, partially blinded, side-by-side comparator study to assess the safety and tolerability, feasibility, and potential added diagnostic and clinical value of using the FerroTrace® and FerroMag Sentinel Lymph Node Mapping (SLNM) System for mapping sentinel lymph nodes (SLNs) in subjects with gastric, gastric-oesophageal junction, and oesophageal cancers, consisting of a safety lead-in phase and an expansion phase.

DETAILED DESCRIPTION:
This is a multi-centre, partially blinded, side-by-side comparator study to assess the safety and tolerability, feasibility, and potential added diagnostic and clinical value of using the FerroTrace® and FerroMag SLNM System for mapping SLNs in subjects with gastric, gastric-oesophageal junction, and oesophageal cancers, consisting of a safety lead-in phase and an expansion phase.

A safety lead-in phase will be adopted to determine the optimal dose for the expansion phase. For the safety lead-in phase, a minimum of 6 eligible subjects will undergo a FerroTrace® injection followed by Research magnetic resonance imaging (MRI) to visualise and assess SLNs. Safety will be monitored for 7 to 14 days, and will include reviews of safety, pharmacokinetics, image quality data from MRI pre and post FerroTrace® injection, and MRI SLN identification feasibility. Dose escalation/de-escalation may be performed using a 3+3 design if required. Upon successful completion of the safety lead-in phase, a dose of FerroTrace® will be selected for use in the expansion phase.

The expansion phase will consist of three cohorts of subjects (gastric, gastric-oesophageal junction, oesophageal cancers). Eligible subjects will undergo a FerroTrace® injection followed by a Research MRI to visualise and assess SLNs. If applicable a post neoadjuvant therapy Research MRI may be performed. The Research MRIs will be blinded to the multi-disciplinary team (MDT). During surgery a comparator product, Indocyanine green (ICG) with a near-infrared camera, will be used to identify fluorescent lymph nodes and in histopathology on ex-vivo specimens a magnetometer (FerroMag) will identify SLNs. The identification and location of all identified SLNs will be recorded, and all will be examined with fine serial sectioning and immunochemistry by pathology.

The study will assess disease free and overall survival and its correlation to histopathology and SLN location.

ELIGIBILITY:
Inclusion Criteria:

* Subject is capable of understanding and has provided written informed consent.
* Subject over 18 years of age and is fit to complete the study in the opinion of the investigator.
* Subject with a previously untreated histopathology confirmed diagnosis of gastric, gastric-oesophageal junction, oesophageal cancer and at the time of enrolment is expected to undergo curative-intent surgery.
* Females of childbearing potential must be willing to use methods of contraception as deemed adequate by the Investigator to be eligible for, and continue participation in, the study.
* In the opinion of the Investigator, the subject can complete the study in compliance with the Investigational Plan and is able to comply with the requirements of the Investigational Plan.
* Subjects with an Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0-2.
* Additional tumour specific inclusion criteria for subjects in expansion cohorts as directed by the Sponsor.

Exclusion Criteria:

* Subject has distant metastasis as detected on CT, PET, ultrasound guided fine needle aspiration (FNA), or cytology prior to enrolment.
* Subject started neoadjuvant therapy before informed consent, or prior to FerroTrace® administration.
* Subject has received a Feraheme® (ferumoxytol) injection within the past 180 days.
* Subject has a known or suspected history of allergies, hypersensitivity, or intolerances as follows:

  1. Iron compounds
  2. Polyacrylamide
  3. Polyethylene glycol (PEG) or has had an anaphylactic reaction to the Pfizer or Moderna COVID vaccines
  4. Iodine compounds
  5. Known or suspected hypersensitivity to FerroTrace®, or to any ingredients of FerroTrace®.
* Subject known to have haemochromatosis.
* Subjects with other known iron metabolism disorder(s) if the Investigator determines the subject is at a higher risk of iron toxicity.
* Subjects who at the time of enrolment are pregnant or lactating, or from the time of enrolment through to 14 days after injection of the study dose are trying to become pregnant, planning to impregnate a partner, or planning to donate sperm.
* Subject has one or more absolute contraindications to MRI scanning as per Investigator judgement.
* Subjects with an estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73m2.
* Subject has inability or unwillingness to comply with all follow-ups through to the end of the study, and/or unwilling to allow review of medical records in accordance with local regulatory requirements at time of consent.
* Investigator determines that the subject is not suitable for study participation for any other reason.
* Subject received an investigational product (IP) within 30 days of FerroTrace® administration unless agreed by the sponsor.
* Subjects have hyperthyroidism or benign thyroid nodules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
SLN detection rate | Up to 14 days post surgery
  SLN detection rate and number of SLNs per subject using MRI and FerroMag following FerroTrace® injection and concordance between MRI and FerroMag
Ultra-staging diagnostic value | Up to 14 days post surgery
  Positive diagnostic value of FerroTrace® SLN mapping and SLN histopathological ultra-staging defined as the number of additional node negative (pN0/ypN0) subjects who are diagnosed with isolated tumor cells (pN0i+/ypN0i+), micro-metastasis (pN1mi/ypN1mi) and node positive (pN1/ypN1) by SLN ultra-staging plus standard of care histopathology versus standard of care histopathology only.
Surgical quality | Up to 14 days post surgery
  Percentage of subjects with an SLN identified on MRI that is/are untreated by radiotherapy or surgery.

SECONDARY OUTCOMES:
Rate of Adverse Events (AEs) | The earlier of 28 days post FerroTrace injection or commencement of neoadjuvant therapy or surgery
  Incidence, nature, severity, and relatedness to FerroMag or FerroTrace® of AEs and Serious Adverse Events (SAEs), changes of laboratory parameters, vital signs, and ECG results per NCI CTCAE v5.0
SLN Location Disease Free Survival | Up to 5 years post surgery
  Disease free survival rates of subjects categorised by SLN location (MRI identified SLNs all treated/removed by radiotherapy/surgery versus some SLNs not treated/removed).
SLN Ultra-staging Disease Free Survival | Up to 5 years post surgery
  Disease free survival rates of subjects categorised by histopathology after SLN ultra-staging.
SLN Location Overall Survival | Up to 5 years post surgery
  Overall survival rates of subjects categorised by SLN location (MRI identified SLNs all treated/removed by radiotherapy/surgery versus some SLNs not treated/removed)
SLN Ultra-staging Overall Survival | Up to 5 years post surgery
  Overall survival rates of subjects categorised by histopathology after SLN ultra-staging

OTHER OUTCOMES:
FerroTrace and ICG Concordance | Up to 14 days post surgery
  Nodal yield of ICG nodal mapping and concordance rate of FerroTrace® identified SLNs versus ICG identified nodes, categorised by subjects' neoadjuvant therapy type if applicable
FerroTrace enhanced MRI Diagnosis | Up to 14 days post surgery
  Specificity and sensitivity of FerroTrace® enhanced MRI in detecting tumour deposits in the SLNs versus CT, positron emission tomography (PET), and standard of care histopathology
FerroTrace enhanced MRI Response | Up to 14 days post surgery
  Specificity and sensitivity of FerroTrace® enhanced MRI in detecting response to neoadjuvant therapy in lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Joe El-Aklouk, Study Director — Ferronova Pty Ltd
Locations (4):
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No